CLINICAL TRIAL: NCT02992327
Title: Biomarker Levels as A Predictor of Concussion Severity OUTcomes (BlacOut)
Acronym: BlacOut
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: A15-085
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Concussion, Mild; Neurocognitive Dysfunction
MeSH Terms: conditions — Brain Concussion; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The laboratory has developed and characterized extensively an antibody that reacts with the SNTF (structural brain protein calpain-cleaved αII-spectrin N-terminal fragment) fragment of aII-spectrin but does not recognize either the intact aII-spectrin or any other fragment of it. The laboratory has used this antibody as a foundation for an ultrasensitive, specific, standardized sandwich immunoassay for measuring trace quantities of SNTF in human serum and plasma in the acute period after brain injury19,27 The method employs state-of-the-art electrochemiluminescence chemistry that is widely used in the clinical diagnostics arena for measuring protein biomarkers in biological fluids.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients age ≥ 8 years of age with a GCS >13 presenting to the emergency department with a diagnosis of concussion.

SUMMARY:
The overall research aim of this pilot study is to determine if the structural brain protein calpain-cleaved αII-spectrin N-terminal fragment (SNTF) can be used as a blood biomarker to accurately identify patients who will have more severe symptoms and reduced neurocognitive functioning after sustaining a concussion. Concussion is also referred to as mild traumatic brain injury (mTBI) in the literature. Both terms will be used interchangeably throughout this application.

DETAILED DESCRIPTION:
The novel aspect of the proposed study relates to the fact that the STNF protein is the first evidence that a biomarker in human blood can help clinicians determine a specific patient's clinical outcome from a concussion. This in turn will help clinicians and concussion specialists with designing treatment protocols very early after the initial injury that could have significant impacts on the health of the patient.

This study has several important benefits to the scientific community. Concussion treatment today is uncertain. Some patients are back to baseline one or two days post injury whereas other patients are experiencing debilitating symptoms for months after the injury. Until the patient begins to report symptoms, the course of treatment cannot be determined. Other biomarkers for concussion diagnosis are being evaluated, but this is the first biomarker to show promise for patient stratification and earlier intervention and treatment for the subset of cases at high risk of suffering brain damage and persisting dysfunction after concussion. Currently, no prognostic method exists for identifying at an early and potentially treatable stage the small subset of concussion sufferers at risk of diffuse axonal injury and persisting brain functional impairment.

ELIGIBILITY:
Inclusion Criteria:

Patient is ≥ 8 years old 2. Ability to enroll within 24 hours of injury 3. Ability to follow-up with patient 30 days following enrollment 4. Concussion by history or physical examination (head injury and symptoms such as headache, nausea, vomiting, dizziness, fatigue, irritability, or poor concentration following the injury) 5. GCS ≥ 13 6. Abbreviated Injury Score (AIS) ≤ 3 7. Plan to be discharged from the emergency department to the outpatient observation unit or to home

Exclusion Criteria:

Non-English speaking 2. Trauma Team Activation (TTA) 3. Abnormal acute intracranial CT/MRI findings 4. Blood alcohol level (> 200 mg/dL) 5. Previous head injury within 30 days of enrollment 6. Pre-existing neurologic disorder associated with cerebral dysfunction and/or cognitive deficit (such as dementia, cerebral palsy, mental retardation, epilepsy, dyslexia) 7. Pre-existing psychiatric disorder (such as bipolar disorder and schizophrenia) as indicated by medical history 8. Planned admission to a hospital inpatient unit

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal volunteers presenting to the emergency department with a diagnosis of concussion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-08-30 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Results of neurocognitive testing | 30 days from index injury
  Neurocognitive testing a 30 days post injury to assess symptom severity
Symptom severity | 30 days post injury
  assay level of SNTF biomarker

SECONDARY OUTCOMES:
SNTF plasma and serum levels | 24 hours, 30 days and 90 days post injury
  SNTF plasma and serum levels measured with 24 hours of injury, at 30 days, at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Sandi Wewerka, MPH, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD